CLINICAL TRIAL: NCT07214311
Title: RETAIN: A Phase 2/3 Randomized, Placebo-Controlled Study to Evaluate the Efficacy of PLG0206 in Prevention of Recurrent Infection in Patients Undergoing Debridement, Antibiotics, and Implant Retention (DAIR) for Treatment of a Periprosthetic Joint Infection (PJI) Following Total Knee Arthroplasty (TKA)
Brief Title: Evaluation of PLG0206 in Prevention of Recurrent Infection in Patients Undergoing Debridement, Antibiotics, and Implant Retention (DAIR) for Treatment of a Periprosthetic Joint Infection (PJI) Following Knee Arthroplasty
Acronym: RETAIN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peptilogics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLG0206-PJI-300
Record Dates: First submitted 2025-09-18; First posted 2025-10-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prosthetic-joint Infection
Keywords: PJI; TKA; DAIR; Joint Infection; Knee Replacement; Prosthetic Joint; Arthroplasty; PLG0206
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLG0206 (Experimental): PLG0206 will be administered as an irrigation solution during DAIR procedure
  Interventions: Drug: PLG0206
- Placebo (Placebo Comparator): Placebo (normal saline) will be administered as an irrigation solution during DAIR procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLG0206 — PLG0206 Solution
  Arms: PLG0206
Drug: Placebo — Placebo
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether the investigational drug PLG0206 can help reduce recurrence of infection in adults who have undergone total knee replacement and are receiving a DAIR (Debridement, Antibiotics, and Implant Retention) surgical procedure to treat a Prosthetic Joint Infection (PJI). The study will also assess the safety of PLG0206 when used as an irrigation solution during the DAIR procedure.

Participants will receive either PLG0206 or a placebo (an inactive substance that looks like the investigational drug), in addition to standard of care treatments. All participants will be monitored for approximately one year following their DAIR procedure.

DETAILED DESCRIPTION:
This study is designed to assess the efficacy and safety of PLG0206 administered intraoperatively by local irrigation to participants undergoing a DAIR procedure for treatment of Prosthetic Joint Infection (PJI) occurring after total knee arthroplasty (TKA), also known as knee joint replacement.

Eligible participants will undergo a DAIR procedure according to the treating hospital's standard of care (SOC). Participant eligibility will be based on clinical and diagnostic assessments, including laboratory results.

Once debridement during DAIR is complete, the Investigator will follow a standardized irrigation protocol, with the final irrigation step being administration of a single dose of blinded study drug (PLG0206 or matching placebo). The study drug will be administered as a single intra-articular irrigation.

Following study drug administration, all participants will receive standard post-operative care per institutional guidelines and will be discharged from the hospital in accordance with local standards. Participants may receive IV/oral antimicrobial therapy, as part of post-operative SOC.

Participants will be monitored for safety and signs of PJI recurrence or persistent infection for 365 days post study drug administration. After hospital discharge, study visits will occur in-clinic on Days 14, 90, and 365, and on Days 30, 180, and 270 via a telephone or virtual visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants age between 18 and <80 years
* Able to provide informed consent, geographically stable, and able to comply with the required follow-up visits
* Suspected or confirmed PJI of the knee
* Well-fixed and positioned prosthesis and good condition of surrounding soft tissue (no sinus tract)
* A single DAIR procedure is indicated as treatment of PJI
* Agree to use contraceptives if of childbearing potential

Exclusion Criteria:

* Loose prosthesis or surgical treatment planned for removal of well-fixed, nonmodular implants
* Anticipated to require antibiotic therapy for >6 months after DAIR procedure
* Infection spread beyond the affected knee joint (e.g., osteomyelitis)
* History of a prior PJI of the affected knee
* Two or more prior revisions in the affected joint
* Epithelialized sinus tract with evidence of communication to the joint or visualization of prosthesis
* Diabetes mellitus and with an A1c ≥9%
* History of malignant disease and having received immunosuppressive therapy, radiation therapy, or chemotherapy within the past year
* Known immunodeficiency (e.g., splenectomy; sickle cell anemia; human immunodeficiency virus [HIV] with recent CD4 count <200 cells/mm3; or primary humoral, bone marrow, or other transplantation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in Treatment Failure Post DAIR | From treatment through 12 months
  Proportion of participants with PJI treatment failure following DAIR

SECONDARY OUTCOMES:
Reduction Rate of PJI-related Surgical Intervention | From treatment through 12 months
  Proportion of participants with PJI requiring a PJI-related surgical intervention following DAIR
Safety of PLG0206 | From treatment through 12 months
  Evaluation of adverse events
Survival | From treatment through 12 months
  Evaluation of PJI-related mortality rate
Efficacy of PLG0206 on Clinical Outcome | At Days 14, 30, 90, 180, 270, and 365
  Evaluate the rate of PJI treatment failure at specific time points
Time to Treatment Failure | From treatment through 12 months
  Evaluation on effect of PLG0206 on time to treatment failure
PJI-related Healthcare Resource Utilization | From treatment through 12 months
  Evaluate the effect of PLG0206 on the need for medical care after post-DAIR procedure discharge
Frequency of PJI-related Surgical Procedures Following DAIR | From treatment through 12 months
  Evaluate the number of surgical procedures for PJI treatment performed after the initial DAIR procedure
Microbiological Efficacy Outcome | From treatment through 12 months
  Evaluate the per-pathogen microbiological response rate following study drug administration
Functional Change Post-DAIR | From Baseline through 9 months
  Evaluate the effect of PLG0206 on the functional change from baseline utilizing the Oxford Knee Scale, where total scores range from 0 (poorest function) to 48 (maximal function)
Immunogenicity of PLG0206 | from Baseline through 12 months
  Evaluation of anti-drug antibodies to PLG0206
Effect of PLG0206 on the inflammatory biomarker C-reactive Protein | Measured at Baseline and Days 14, 90, and 365
  Evaluate the difference between the PLG0206 and placebo groups in normalization of C-reactive protein levels post treatment
Maximum Plasma Concentration (Cmax) of PLG0206 | From Baseline through Day 3
Time to Maximum Plasma Concentration (Tmax) of PLG0206 | Baseline through Day 3
Half-life of PLG0206 in Plasma | Baseline through Day 3
Area Under the Concentration-time Curve Through Last Quantifiable Concentration | From time O (pre-dose) through last quantifiable result; last protocol specified time-point is Day 3
  Characterization of systemic PK of PLG0206
Area Under the Concentration-time Curve Through Infinity | From time O (pre-dose) to infinity [AUCinf]; last protocol specified time-point is Day 3
  Characterization of systemic PK of PLG0206
Concentration of PLG0206 in Irrigation Solution | Measured at Study Day 1 at end of study drug exposure
  Concentration of PLG0206 in irrigation solution at the end of study drug exposure

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Clinical Trial Site, Tamarac, Florida
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Morgantown, West Virginia